CLINICAL TRIAL: NCT06337383
Title: Study of the Prevalence of Autistic Traits in Angelman Syndrome, the Correlation With Cognitive Level, Epilepsy, With Socio-communication Skills and Parenting Styles
Brief Title: Study of the Prevalence of Autistic Traits in Angelman Syndrome
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 12.2021 ANGELMAN
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational cross-sectional study is to establish the prevalence of autism spectrum disorder in children and adolescents with Angelman syndrome. The main questions it aims to answer are:

* which clinical variables differentiate AS patients with and without Autism Spectrum Disorder between genetics, epilepsy, pharmacotherapy, behavioural problems, parenting style and parents' perceived stress.
* which clinical variables differentiate parenting styles and levels of perceived stress.

Data from neuropsychological, speech therapy and physiotherapeutic assessments are collected during regular clinical follow-ups, regarding: cognitive development ("Bayely Scales of Infant Development-III", Cognitive Scale) and adaptive behaviour; Autism and Autism Spectrum Disorder ("Autism Diagnostic Observational Schedule-2"); parental stress and parenting styles; social-communicative skills; motor development.

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed diagnosis of Angelman Syndrome
* chronological age between 4-15 years

Exclusion Criteria:

* genetic examination pending report
* mental age lower than 12 months
* brain injury acquired in the peri- or postnatal period

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants are recruited at I.R.C.C.S. "E. Medea", in Conegliano (Italian referral centre for Anelman Syndrome) in collaboration with Or.S.A (the Italian organisation for the syndrome).
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Total score of the Autism Diagnostic Observation Schedule -2 (ADOS-2), Module 1, | Once at recruitment
  The ADOS-2 consists of different semi-structured standard situations that induce communication, social interaction and imaginative play and that is considered a gold standard in autism assessment; Module 1, that does not require the use of speech, is employed.
  In particular, our outcome of interest is the "Total score", given by the sum of the "Communication and Reciprocal Social Interactions" and the "Stereotyped Behaviors and Restricted Interests" raw scores. Higher scores correspond to a greater presence of autistic features (min:0; max:28; cut-off for autism spectrum disorder:11; cut-off for autism disorder:16).

SECONDARY OUTCOMES:
Age-equivalent score at the Cognitive Scale of the Bayley Scales of Infant Development - 3rd version (Bayley-III) | Once at recruitment
  The Bayley-III Cognitive Scale is used to assess cognitive level. In particular, age-equivalent scores are considered (min: 1 months; max: 42 months).
Total Stress score at the Parent Stress Index - 4th edition (PSI-4) questionnaire | Once at recruitment
  PSI-4 is a standardised parent self-report instrument to explore perceived stress in their role and therefore to identify situations at risk of dysfunctional parent-child system. It is composed of two subscales: the child domain, that identifies six child characteristics, and the parent domain, that describes seven stressors related to parent and family characteristics. Our outcome of interest is the Total Stress score, given by the sum of the scores obtained at the "Child domain" and the "Parent domain".
  Higher scores correspond to a greater level of parental stress.
Global score at the Aberrant Behaviour Checklist (ABC) | Once at recruitment
  The ABC is a questionnaire that measures psychiatric symptoms and behavioural disturbance in individuals with severe or very severe intellectual disability across 5 domains: irritability, agitation and crying; lethargy/social withdrawal; stereotypic behaviour; hyperactivity/noncompliance; inappropriate speech. It is useful to assess the possible effects of medications or other treatments. In particular is considered the Global score, obtained from the sum of the scores at each subscale (min: 0; max: 171; higher scores correspond to a greater level of behavioural problems).
Total Raw score at the Social Communication Questionnaire - Current version(SCQ) | Once at recruitment
  Children's communication, social and interpersonal skills are indirectly investigated through the Social Communication Questionnaire- Current version. It screens for characteristics associated with Autism (cut-off: 22) and Autism Spectrum Disorder (cut-off: 15) such as social interaction, communication and repetitive behaviour, considering the last three months (min: 0; max: 33).

CONTACTS AND LOCATIONS:
Overall Officials: Martina Baggio, Principal Investigator — Scientific Institute IRCCS E. Medea, Epilepsy Unit, Conegliano 31015, Italy
Locations (1):
- I.R.C.C.S. "E.Medea", Conegliano, Treviso, Italy